CLINICAL TRIAL: NCT06368388
Title: Bacteriophage Therapy for Difficult-to-treat Infections: the Implementation of a Multidisciplinary Phage Task Force
Acronym: PHAGEFORCE
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S64854
Record Dates: First submitted 2024-04-04; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Musculoskeletal Infection; Chronic Rhinosinusitis (Diagnosis); Sepsis; Pulmonary Infection; Hidradenitis Suppurativa
Keywords: Bacteriophage therapy; Personalized treatment; Difficult-to-treat infection
MeSH Terms: conditions — Disease; Sepsis; Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phage treated group: Solely depending on the susceptibility of the isolates against the available phages (phagogram) the CBL will decide if the patient can be included in the phage treated group or the control group. Patients in the phage treated group will receive phage therapy according to the medical indication (local for musculoskeletal infections, hidradenitis suppurativa and CRS, through inhalation for pulmonary infections, intravenous for sepsis) on top of (surgical/antimicrobial) standard treatment.
  Interventions: Other: Prospective data collection
- Control group: Patients for whom the isolated pathogens are not susceptible to the available phages are included in the control group. These patients receive standard (non-curative) surgical/antimicrobial treatment.
  Interventions: Other: Prospective data collection

INTERVENTIONS:
Other: Prospective data collection — Prospective data collection prior to, during and after phage treatment.
  Groups: Phage treated group
Other: Prospective data collection — Prospective data collection prior to, during and after standard infection treatment.
  Groups: Control group

SUMMARY:
PHAGEFORCE is a prospective, observational registry study. The University Hospitals Leuven has approved the application of phage therapy as standard-of-care only in patients for whom no curative treatment alternatives (antibiotic and/or surgical) are available ('last-resort cases'). A multidisciplinary phage task force, referred to as the Coordination group for Bacteriophage therapy Leuven (CBL) was set up. The CBL screens patients with difficult-to-treat infections, evaluates who could benefit from phage therapy and sets up the treatment protocol. With this study, the CBL aims to gain insight in the safety and efficacy of phage therapy by integrating and optimizing phage therapy in five distinct medical disciplines (with distinct routes of administration), facilitating long-term follow-up of patients. Furthermore, this study will gain insight in the biodistribution and exact mechanisms of action of phage therapy and thus be able to provide standardized guidelines for each patient population and route of administration.

DETAILED DESCRIPTION:
Patients with difficult-to-treat musculoskeletal infections, chronic rhinosinusitis, sepsis, pulmonary infections associated with cystic fibrosis or bronchiectasis, or hidradenitis suppurativa, for whom no standard (curative) treatment options are available, are eligible for phage therapy. Patient eligibility is evaluated by the Coordination group for Bacteriophage therapy Leuven. If phages are available against the isolated bacterial species and the patient is found eligible for phage therapy, a phagogram is performed. Solely based on the results of the phagogram, the patient is either included in the phage treated or control group (standard (non-curative) treatment). In both cases, data is collected using REDCap.

ELIGIBILITY:
Inclusion Criteria:

All patients:

* Diagnosed with a musculoskeletal infection or chronic rhinosinusitis or sepsis or lung infection (CF/Bx) or hidradenitis suppurativa, and
* For whom all previous treatments (surgical and antibiotic) have failed or for whom no other treatment options are available (i.e., last resort cases, based on the assessment of the CBL), for example in case of bacterial resistance. And
* Of whom the pathogen causative for the infection is one for which phages are available in the phage bank, and
* Who have given informed consent to have their data collected in a patient registry

Exclusion Criteria:

All patients:

* With an infectious disease other than those mentioned above, and/or
* For whom standard treatment alternatives are still available. And/or
* Of whom the pathogen causative for the infection is not one for which phages are available in the phage bank. And/or
* Who refused to give their informed consent

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a musculoskeletal infection or sepsis or chronic rhinosinusitis or pulmonary infection (associated with bronchiectasis or cystic fibrosis) or hidradenitis suppurativa for whom all previous treatments (anti-inflammatory/antibiotic/surgical) have failed or are likely to fail, or for whom no other treatments are available (i.e. in case of antibiotic resistance).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease free period | 1 year after treatment
Bacterial eradication | 3 months after treatment
  specific to sepsis patients, evaluated by negative hemocultures

SECONDARY OUTCOMES:
PROMIS global health (patient-reported outcome measurement information system) | until 1 year after treatment
  specific to musculoskeletal infections, chronic rhinosinusitis and pulmonary infections; higher scores mean better outcome
PROMIS (patient-reported outcome measurement information system) physical function | until 1 year after treatment
  specific to musculoskeletal infections (higher scores mean better outcome)
PROMIS (patient-reported outcome measurement information system) pain interference | until 1 year after treatment
  specific to musculoskeletal infections (higher scores mean worse outcome)
Sino-nasal outcome test (SNOT)-22 | until 1 year after treatment
  specific to chronic rhinosinusitis, lower scores mean a better outcome
Visual Analogue Scale (VAS) score | until 1 year after treatment
  specific to chronic rhinosinusitis and hidradenitis suppurativa, higher scores mean more pain
Cystic fibrosis questionnaire (CF-Q-R) | until 1 year after treatment
  specific to pulmonary infections, higher scores mean better quality of life
Dermatology Life Quality Index (DLQI) | until 1 year after treatment
  specific to hidradenitis suppurativa, higher scores mean worse outcome (impaired quality of life)
Hidradenitis Suppurativa Quality of Life (HiSQoL) | until 1 year after treatment
  specific to hidradenitis suppurativa, higher scores indicate a higher level of symptomatology (worse outcomes)

OTHER OUTCOMES:
Rate of exacerbations | until 12 months after treatment
  specific to pulmonary infections
Abscess and inflammatory nodule (AN) count with Hidradenitis suppurativa Clinical Response (HiSCR) | until 3 months after treatment
  specific to hidradenitis suppurativa. At least a 50% reduction from baseline in the total AN count, with no increase from baseline in abscess or draining tunnel count
Lund-Mackay CT score | until 3 months after treatment
  specific to chronic rhinosinusitis, higher scores mean more occlusion
Lund Kennedy endoscopy score | until 3 months after treatment
  specific to chronic rhinosinusitis, higher scores mean more occlusion
Modified Davos score | until 3 months after treatment
  specific to chronic rhinosinusitis, higher scores mean more occlusion

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Background] Onsea J, Uyttebroek S, Chen B, Wagemans J, Lood C, Van Gerven L, Spriet I, Devolder D, Debaveye Y, Depypere M, Dupont L, De Munter P, Peetermans WE, van Noort V, Merabishvili M, Pirnay JP, Lavigne R, Metsemakers WJ. Bacteriophage Therapy for Difficult-to-Treat Infections: The Implementation of a Multidisciplinary Phage Task Force (The PHAGEFORCE Study Protocol). Viruses. 2021 Aug 5;13(8):1543. doi: 10.3390/v13081543. PMID 34452408